CLINICAL TRIAL: NCT07011823
Title: Phase II Trial of Immunochemotherapy and Partial Breast Irradiation in Early TNBC With Immune-cold Tumor Environment (KEY-MELT)
Brief Title: Immune-checkpoint Blockade After Partial Breast Irradiation by Pembrolizumab in Early TNBC
Acronym: KEY-MELT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2025-0070
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Triple-Negative Breast Neoplasm
Keywords: Immune-cold microenvironment; Triple-negative breast cancer; Partial Breast Irradiation; Pembrolizumab; KeyNote-522; Immunochemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunochemotherapy including pembrolizumab after partial breast-irradiation (Experimental): First, 8Gy partial breast irradiation will be delivered in immune-cold triple-negative breast cancer (TNBC) confirmed by PD-L1 and TILs.
  Sequentially, standard neoadjuvant chemotherapy for triple-negative breast cancer including pembrolizumab, paclitaxel, carboplatin, doxorubicin, and cyclophosphamide (KeyNote-522 regimen) will be administered, followed by surgical treatment.
  Interventions: Radiation: Partial breast-irradiation

INTERVENTIONS:
Radiation: Partial breast-irradiation — First, 8Gy partial breast irradiation will be delivered in immune-cold triple-negative breast cancer (TNBC) confirmed by PD-L1 and TILs.
  Sequentially, standard neoadjuvant chemotherapy for triple-negative breast cancer including pembrolizumab, paclitaxel, carboplatin, doxorubicin, and cyclophosphamide (KeyNote-522 regimen) will be administered, followed by surgical treatment.

SUMMARY:
A single-arm, single-institution study to induce phenotypic changes in the tumor microenvironment by delivering 8Gy partial breast irradiation in immune-cold triple-negative breast cancer confirmed by PD-L1 and TILs. Additional tissue biopsy will be performed following radiation therapy. Subsequently, neoadjuvant chemotherapy including Pembrolizumab will be administered to evaluate whether pathological complete response rates are improved.

DETAILED DESCRIPTION:
A single-arm, single-institution study to induce phenotypic changes in the tumor microenvironment by delivering 8Gy partial breast irradiation in immune-cold triple-negative breast cancer confirmed by PD-L1 and TILs. Additional tissue biopsy will be performed following radiation therapy.

Subsequently, under the supervision and management of breast surgery and medical oncology research teams, standard neoadjuvant chemotherapy for triple-negative breast cancer including pembrolizumab, paclitaxel, carboplatin, doxorubicin, and cyclophosphamide (KeyNote-522 regimen) will be administered, followed by surgical treatment.

Pathological complete response status in surgical specimens will be confirmed and reported by the pathologist.

Pathological examination and spatial multiplex analysis will be performed on biopsy and surgical specimens to explore biomarkers with significant changes.

As secondary end-points, disease-free survival and overall survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients aged 20 years or older with clinical stage IIA or higher on imaging studies
* Patients with triple-negative breast cancer confirmed on tissue biopsy
* Cold immune tumor environment with tumor-infiltrating lymphocytes (TILs) <30% and PD-L1 Combined Positive Score (CPS) <10 on immunohistochemical staining of biopsy specimens
* Patients with no prior history of breast cancer
* Patients with no prior history of chemotherapy or radiation therapy
* Patients scheduled to receive partial breast irradiation
* Patients with ECOG performance status of 0-2
* Patients who voluntarily signed the informed consent form for study participation

Exclusion Criteria:

* Patients with non-triple-negative breast cancer on tissue biopsy
* Patients scheduled for surgery without neoadjuvant chemotherapy
* Patients with TILs ≥30% or PD-L1 CPS ≥10 on immunohistochemical staining of biopsy specimens (immune-hot tumor)
* Patients with recurrent breast cancer or de novo stage IV disease
* Patients who have previously received chemotherapy and/or radiation therapy to the ipsilateral breast and chest prior to study participation
* Patients unable to receive neoadjuvant chemotherapy and Pembrolizumab
* Vulnerable research subjects who are unable to participate voluntarily in the study due to physical/mental disabilities

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Within 3 weeks after surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung Gwe Ahn, Principal Investigator — M.D.,Ph.D.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schmid P, Cortes J, Dent R, McArthur H, Pusztai L, Kummel S, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Im SA, Untch M, Fasching PA, Mouret-Reynier MA, Foukakis T, Ferreira M, Cardoso F, Zhou X, Karantza V, Tryfonidis K, Aktan G, O'Shaughnessy J; KEYNOTE-522 Investigators. Overall Survival with Pembrolizumab in Early-Stage Triple-Negative Breast Cancer. N Engl J Med. 2024 Nov 28;391(21):1981-1991. doi: 10.1056/NEJMoa2409932. Epub 2024 Sep 15. PMID 39282906